CLINICAL TRIAL: NCT00047944
Title: Neural Circuitry and Risk for Depression in Adolescents: A Study Using Functional Magnetic Resonance Imaging
Brief Title: MRI Study of Brain Activity and Risk for Depression in Adolescents
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030014; 03-M-0014
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-10-27

CONDITIONS: Involutional Depression; Anxiety Disorders
Keywords: Attention; Emotion; Amygdala; Prefrontal Cortex; Facial Expression; Magnetic Resonance Imaging; fMRI; Depression; Anxiety; Adolescence; Children
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Facial Expression; Depression

SUMMARY:
Anxiety in children of parents with major depressive disorder (MDD) poses a particularly high risk for later-life MDD. In adults, MDD involves dysfunction in prefrontal brain regions that regulate attention to emotional stimuli. These abnormalities: i) have been found primarily in adults with specific familial forms of MDD; ii) persist after recovery from MDD, and iii) relate to anxiety. These findings raise the possibility that risk for MDD is tied to dysfunction in prefrontal regions involved in regulation of emotion, which possibly manifests as early-life anxiety. If this possibility were confirmed in never-depressed adolescents at high risk for MDD, the findings would provide key insights into the developmental neurobiology of MDD. The goal of this protocol is to study the neural substrate of risk for MDD in young people. This protocol tests the hypothesis that adolescents at high risk for MDD by virtue of childhood anxiety and parental history of MDD exhibit dysfunction in prefrontal cortex and amygdala, regions involved in emotion regulation. This goal will be accomplished through fMRI studies of emotion regulation in high and low-risk adolescents.

For this research, at-risk adolescents will be recruited from participants in an NIMH-funded extramural study at New York University (NYU) examining the biology of risk for anxiety and depressive disorders. Over a three-year period, 45 high-risk probands and 60 low-risk comparisons will be studied, including 20 comparisons from the NYU sample and 40 from the Washington DC metropolitan area. In the present protocol, to be conducted at NIH, subjects will undergo volumetric MRI scans to assess structural abnormalities in the prefrontal cortex and medial temporal lobe. They will complete a series of four out-of-scanner cognitive tasks and two fMRI-based cognitive tasks that measure modulation of attention to emotional stimuli. The fMRI tasks are hypothesized to differentially engage the prefrontal cortex and amygdala in low vs. high risk subjects. These tasks will be used to test the hypothesis that at-risk individuals exhibit enhanced amygdala and reduced prefrontal activation on the fMRI emotion/attention tasks.

DETAILED DESCRIPTION:
Parental history of major depressive disorder poses a particularly high risk for later-life MDD. In adults, MDD involves dysfunction in subcortical brain regions related to emotional responsiveness, such as the amygdala, and in cortical brain regions that interface cognitive and emotional processes. These abnormalities: i) have been found primarily in adults with specific familial forms of MDD; ii) persist after recovery from MDD, and iii) relate to anxiety. These findings raise the possibility that risk for MDD is tied to dysfunction in emotional circuits themselves or in prefrontal regions involved in regulation of emotion. If this possibility were confirmed in never-depressed adolescents at high risk for MDD, the findings would provide key insights into the developmental neurobiology of MDD. The goal of this protocol is to study the neural substrate of risk for MDD in young people. This protocol tests the hypothesis that adolescents at high risk for MDD by virtue of parental history of MDD exhibit dysfunction in prefrontal cortex, amygdala, and other subcortical regions involved in emotion and emotion regulation. This goal will be accomplished through fMRI studies of edmotion provocation in high and low-risk adolescents.

For this research, at-risk adolescents will be recruited from participants in NIMH-funded extramural studies at New York University, Brown University, and Columbia University examining the biology of risk for anxiety and depressive disorders. Over a three-year period, data on each measure of interest will be obtained in 100 high-risk probands and 100 low-risk comparisons. In addition, a sub-set of parents of these adolescents (n=100) also will be studied using identical procedures. In the present protocol, to be conducted at NIH, subjects will undergo volumetric MRI scans to assess structural abnormalities in the prefrontal cortex and medial temporal lobe. They will complete a series of out-of-scanner cognitive tasks and fMRI-based cognitive tasks. Two of these tasks measure modulation of attention to emotional stimuli; the third task measures engagement of temporal and prefrontal regions during social interactions. For these types of tasks, prior studies in adolescents with ongoing mood and anxiety disorders demonstrate hypothesized abnormalities in brain engagement. The current study is designed to examine the degree to which comparable findings emerge in unaffected adolescents at risk for mood and anxiety disorders.

ELIGIBILITY:
* OFFSPRING SUBJECTS - INCLUSION CRITERIA:

Age: 10-30.

Can give consent/assent. Parents will provide consent for all minors.

All subjects will have IQ greater than 80.

High risk Psychopathology: Offspring of adults with a history of MDD.

Low risk Psychopathology: Offspring of adults with no history of MDD and low developmental levels of emotion dysregulation. Subjects born to parents with only anxiety disorders will be included in this group.

OFFSPRING SUBJECTS - EXCLUSION CRITERIA:

Any medical condition that increases risk for MRI (e.g. pacemaker, metallic foreign body in eye).

Pregnancy:

Both groups: All subjects will be free of current impairing affective disorders, separation anxiety disorder, social anxiety disorder, panic disorder, generalized anxiety disorder, PTSD, ADHD, as well as lifetime history of substance dependence, psychosis, pervasive developmental disorder, major affective disorder, obsessive compulsive disorder, conduct disorder, anorexia. All subjects will be born to parents with no history of schizophrenia or bipolar disorder.

PARENT SUBJECTS - INCLUSION CRITERIA:

Age: 18-55

Can give consent/assent

Offspring: All subjects will have offspring participating in this same protocol.

Have an IQ greater than 80

Past history of MDD

No lifetime history of MDD

ADULT SUBJECTS - EXCLUSION CRITERIA:

Any medical condition that increases risk for MRI (e.g. pacemaker, metallic foreign body in eye)

Pregnancy:

Both groups: All subjects will be free of current significantly impairing affective disorders, psychotropic medications, as well as lifetime history of substance dependence, psychosis, conduct disorder, or anorexia.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2002-10-12; Study Completion 2016-10-27

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Drevets WC, Ongur D, Price JL. Neuroimaging abnormalities in the subgenual prefrontal cortex: implications for the pathophysiology of familial mood disorders. Mol Psychiatry. 1998 May;3(3):220-6, 190-1. doi: 10.1038/sj.mp.4000370. PMID 9672897
- [Background] Drevets WC. Neuroimaging and neuropathological studies of depression: implications for the cognitive-emotional features of mood disorders. Curr Opin Neurobiol. 2001 Apr;11(2):240-9. doi: 10.1016/s0959-4388(00)00203-8. PMID 11301246
- [Background] Drevets WC. Neuroimaging studies of mood disorders. Biol Psychiatry. 2000 Oct 15;48(8):813-29. doi: 10.1016/s0006-3223(00)01020-9. PMID 11063977